CLINICAL TRIAL: NCT07124221
Title: A Randomized, Double-blind, Double-dummy, Positive Controlled, Multicenter Clinical Study to Evaluate the Efficacy and Safety of Cabergoline Tablets Compared With Bromocriptine Mesylate Tablets in Female Patients With Hyperprolactinemia
Brief Title: A Phase III Clinical Study of Cabergoline Tablets Compared With Bromocriptine Mesylate Tablets
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci127-301
Record Dates: First submitted 2025-08-03; First posted 2025-08-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hyperprolactinemia
MeSH Terms: conditions — Hyperprolactinemia | interventions — Cabergoline; Bromocriptine

STUDY DESIGN:
Intervention Model Description: Cabergoline tablets compared with Bromocriptine mesylate tablets
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabergoline tablets (Experimental): 191subjects
  Interventions: Drug: Cabergoline tablets
- Bromocriptine mesylate tablets (Active Comparator): 191subjects
  Interventions: Drug: Bromocriptine mesylate tablets

INTERVENTIONS:
Drug: Cabergoline tablets — Cabergoline tablets will be administered for 14 weeks.The allowed dose range is from 0.25 mg (1 tablet) QW to 1mg (4 tablets) QW. Dosage adjustments are made based on the serum PRL level.
  Arms: Cabergoline tablets
Drug: Bromocriptine mesylate tablets — Bromocriptine mesylate tablets was administered for 14 weeks.The dose is 1.25 mg (0.5 tablet) QD to 7.5mg 3 tablets) QD. Dosage adjustments are made based on the serum PRL level.
  Arms: Bromocriptine mesylate tablets

SUMMARY:
A Phase III clinical study evaluating the efficacy and safety of cabergoline tablets versus bromocriptine mesylate tablets in patients with hyperprolactinemia

DETAILED DESCRIPTION:
A randomized, double-blind, double-dummy, active controlled, multicenter Phase III clinical study to evaluate the efficacy and safety of Cabergoline tablets compared with Bromocriptine mesylate tablets in female patients with hyperprolactinemia

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45 at the time of signing the ICF;
* Clinically diagnosed hyperprolactinemia, with or without pituitary PRL tumor;
* Agree to and abide by the adoption of effective contraceptive measures during the study period (from signing the ICF to 4 weeks after the last administration of the investigational drug);
* voluntarily signed the ICF, could understand and abide by the requirements of this research protocol, and were followed up regularly and on time.

Exclusion Criteria:

* Women who are pregnant or breastfeeding;
* Those who have previously received carbergoline treatment or radiotherapy, or have a history of allergy to ergol preparations or their derivatives;
* The presence of other types or mixed pituitary tumors；
* hyperprolactinemia syndrome caused by hypothalamic or other intracranial lesions；
* hyperprolactinemia syndrome caused by other systemic diseases;
* Laboratory tests during the screening period meet any of the following conditions:

  1. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times ULN, or total bilirubin (TBIL) > 1.5 times ULN, or serum creatinine (Cr) or UREA (UREA)/urea nitrogen (BUN) > 2 times ULN;
  2. Those who are positive for hepatitis B surface antigen, hepatitis C antibody, HIV antibody and Treponema pallidum antibody;
  3. Hyperprolactinemia: Screening tests show that the PRL recovery rate is less than 40%;
* Those who have received ovulation-inducing agents, drugs that may cause an increase in PRL or other prohibited combination drugs within 4 weeks prior to screening;
* The patients not suitable for participating in this clinical study due to other reasons.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 382 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-11-21 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects whose serum PRL levels returned to normal | 14 weeks

SECONDARY OUTCOMES:
The percentage of subjects whose ovulatory cycles resumed | 14 weeks
The percentage of subjects whose galactorrhea disappeared | 14 weeks
The percentage of subjects with pituitary PRL tumor shrinkage | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China